CLINICAL TRIAL: NCT00432822
Title: Double-Blind, Placebo Controlled, Multicentre Study With an Open Label Extension to Evaluate the Efficacy and Safety of Tetrahydrobiopterin (BH4) in Children and Adolescents With Hyperphenylalaninemia Caused by Phenylalanine Hydroxylase Deficiency
Brief Title: Long-Term Tetrahydrobiopterin Treatment in PKU Patients of 0-18 Years - Study on Phenylalanine Tolerance and Safety
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Orphanetics Pharma Entwicklungs GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BH4/III/05/001; EudraCT Number: 2006-000648-15
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Phenylalanine Hydroxylase Deficiencies
Keywords: phenylketonuria; phenylalanine hydroxylase deficiency; BH4; responsive; tetrahydrobiopterin; newborns; infants; children; adolescents
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: tetrahydrobiopterin (BH4)

SUMMARY:
The aim of the study is to confirm the efficacy and safety of BH4 in the treatment of hyperphenylalaninemia caused by phenylalanine hydroxylase deficiency in patients responsive to BH4. The primary objective is to assess the effect of BH4 on phenylalanine tolerance compared to placebo under optimal blood phenylalanine control and to demonstrate safety in 12 months long-term treatment. Additionally population PK will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, aged 0-18 years
* Phenylalanine-4-hydroxylase (PAH) deficiency shown by mutation analysis
* Blood phenylalanine concentration in the target range under dietary treatment
* Written consent of a parent or legal representative
* Assumed availability within the period of study participation
* Patients/parents willing and able to follow the recommended diet
* Use of an effective method of contraception in female patients of child bearing potential

Exclusion Criteria:

* BH4-deficiency due to genetic disorders in biosynthesis or recycling of BH4
* History or current evidence of poor diet compliance
* History or current evidence of clinically relevant allergic or idiosyncratic reactions to drugs or food
* History of allergic reactions to BH4 or its excipients
* Positive pregnancy test (ß-HCG in serum) and lactating females
* Participation in other drug trials within the last 30 days before start for the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)

PRIMARY OUTCOMES:
dietary phenylalanine tolerance
safety

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Superti-Furga, Prof., Principal Investigator — Centre for Pediatrics and Adolescent Medicine, University of Freiburg, Freiburg, Germany

REFERENCES:
- [Background] Muntau AC, Roschinger W, Habich M, Demmelmair H, Hoffmann B, Sommerhoff CP, Roscher AA. Tetrahydrobiopterin as an alternative treatment for mild phenylketonuria. N Engl J Med. 2002 Dec 26;347(26):2122-32. doi: 10.1056/NEJMoa021654. PMID 12501224